CLINICAL TRIAL: NCT07022860
Title: Radiographic Assessment of the Effects of Platelet-Rich Fibrin on Socket Preservation: A Case-Control Study
Brief Title: Study on Platelet-Rich Fibrin for Preserving Jawbone After Tooth Extraction Using CBCT Imaging in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zahedan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Alireza Ranjbaran, Periodontics Resident, Zahedan University of Medical Sciences
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: IR.ZAUMS.REC.1403.379
Record Dates: First submitted 2025-06-07; First posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Socket Preservation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Split-Mouth PRF Arm (Experimental): Each participant will have two symmetrical tooth extractions. One socket will be randomly assigned to receive platelet-rich fibrin (PRF), and the contralateral socket will serve as a control, healing naturally without any graft material. This split-mouth design allows each participant to act as their own control. Radiographic assessments using cone-beam computed tomography (CBCT) will be conducted at baseline and 3 months to measure bone height, ridge width, and socket fill.
  Interventions: Biological: Platelet-rich fibrin (PRF)
- Split-Mouth Control Arm (No Intervention): Each participant will have two symmetrical tooth extractions. One socket will be randomly assigned to receive platelet-rich fibrin (PRF), and the contralateral socket will serve as a control, healing naturally without any graft material. This split-mouth design allows each participant to act as their own control. Radiographic assessments using cone-beam computed tomography (CBCT) will be conducted at baseline and 3 months to measure bone height, ridge width, and socket fill.

INTERVENTIONS:
Biological: Platelet-rich fibrin (PRF) — Platelet-rich fibrin (PRF) is an autologous blood-derived material prepared by centrifuging the participant's venous blood without anticoagulants. The PRF clot is then compressed into a membrane and inserted into the extraction socket. It serves as a scaffold rich in platelets and growth factors to support bone regeneration and healing.
  Arms: Split-Mouth PRF Arm

SUMMARY:
The goal of this clinical trial is to learn if platelet-rich fibrin (PRF), a substance made from a person's own blood, helps preserve the bone in the jaw after tooth extraction in adults. The main questions it aims to answer are:

Does PRF help reduce the loss of bone height after tooth removal? Does PRF improve how much of the socket fills with new bone?

Researchers will compare extraction sites treated with PRF to untreated sites in the same person to see if PRF helps preserve more bone.

Participants will:

Have two teeth removed on opposite sides of the mouth Receive PRF in one socket, while the other socket is left to heal naturally Undergo 3D X-ray scans (CBCT) right after extraction and again 3 months later

This study will help researchers understand if using PRF alone can improve healing and reduce bone loss after tooth extraction.

ELIGIBILITY:
Inclusion Criteria:

Participants were eligible for inclusion if they met the following criteria:

* Age ≥ 18 years
* Smoking fewer than 10 cigarettes per day
* Presence of adequate bony support (≥ 60%)
* Indications for bilateral tooth extraction
* Patients classified as ASA I or II (American Society of Anesthesiologists).
* No systemic conditions known to impair healing, including the following:

  * Use of bisphosphonates
  * Anticoagulant or antiplatelet therapy
  * History of head and neck radiotherapy
  * Chronic use of NSAIDs or corticosteroids

Exclusion Criteria:

Patients were excluded if they met any of the following conditions:

* ASA classification III or IV
* Pregnancy or lactation
* Presence of active infection at the surgical site or need for medications beyond standard analgesics
* Presence of chronic lesions at the extraction site (patients requiring curettage of the lesion were included; those with acute infection requiring antibiotics were excluded).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2024-09-21 (Actual); Primary Completion 2025-01-18 (Actual); Study Completion 2025-01-18 (Actual)

PRIMARY OUTCOMES:
Change in Vertical Ridge Height from Baseline to 3 Months Post-Extraction as Measured by Cone-Beam Computed Tomography (CBCT) | Immediately post-extraction (baseline) and at 3 months post-extraction
  Vertical ridge height was measured using cone-beam computed tomography (CBCT) at two time points: immediately after tooth extraction (baseline) and at 3 months post-extraction. Measurements were taken from the crest of the alveolar ridge to the apex of the extraction socket on both the buccal and lingual sides. The difference in ridge height between the two time points represents the amount of vertical bone loss. A smaller change indicates better preservation of ridge height. The measurements were performed by a blinded radiologist using standardized 1 mm slice thickness and reference lines drawn from the socket apex to the ridge crest.

SECONDARY OUTCOMES:
Change in Horizontal Ridge Width at 1 mm, 3 mm, and 5 mm Apical to the Crest from Baseline to 3 Months Post-Extraction Measured by CBCT | Immediately post-extraction (baseline) and at 3 months post-extraction
  Horizontal ridge width was measured at 1 mm, 3 mm, and 5 mm below the lingual/palatal crest using cone-beam computed tomography (CBCT). The change in width between baseline and 3 months post-extraction was calculated. Smaller changes indicate better preservation of ridge width. Measurements were made using standardized reference lines and a slice thickness of 1 mm.
Percentage of Socket Fill at 3 Months Post-Extraction as Measured by CBCT | 3 months post-extraction
  The percentage of socket fill was determined using CBCT imaging at 3 months post-extraction. Socket fill refers to the amount of mineralized bone formation within the extraction site. A higher percentage indicates greater bone regeneration. A blinded radiologist performed all measurements using pre-defined reference points and standardized protocols.

CONTACTS AND LOCATIONS:
Locations (1):
- Zahedan University of Medical Sciences, Zahedan, Sistan & Balouchestan, Iran

IPD SHARING:
Plan to Share IPD: Yes
Individual de-identified participant data (IPD), study protocol, statistical analysis plan, informed consent form, and clinical study report will be made available to qualified researchers after study completion and publication of the main article. Access will be granted upon reasonable request through written communication with the corresponding author and will be limited to research purposes. Data will be available for at least five years following publication.
Supporting Information: Study Protocol, SAP, ICF, CSR